CLINICAL TRIAL: NCT02354443
Title: A Phase 1 Trial of a Single ProHema® CB Product as Part of Single Cord Blood Unit Transplant After Busulfan/Cyclophosphamide/ATG Conditioning for Pediatric Patients With Inherited Metabolic Disorders
Brief Title: A Trial of a Single ProHema-CB Product Transplant in Pediatric Patients With Inherited Metabolic Disorders
Acronym: PROVIDE
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision
Sponsor: Fate Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FT1050-05
Record Dates: First submitted 2015-01-16; First posted 2015-02-03 (Estimated); Results first posted 2018-10-10 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-02

CONDITIONS: Metabolic Disorders
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ProHema-CB (Experimental): ProHema-CB represents Ex Vivo Modulated Human Cord Blood Cells. Each subject will receive one administration of ProHema-CB unit transplant.
  Interventions: Biological: ProHema-CB Transplant

INTERVENTIONS:
Biological: ProHema-CB Transplant — ProHema-CB, the cellular product, represents the cell populations contained within a human UCB unit after modulation on the day of transplantation by an ex vivo incubation process with the prostaglandin derivative, 16,16-dimethyl prostaglandin E2 (also referred to as FT1050). The cell populations include hematopoietic stem and progenitor cells.

SUMMARY:
The purpose of this study is to describe the safety profile of ProHema-CB as part of a single cord blood unit transplant after a myeloablative conditioning regimen in pediatric patients with inherited metabolic disorders. The safety profile will primarily be assessed by neutrophil engraftment.

DETAILED DESCRIPTION:
This study is an open-label trial of the safety of a single cord blood transplant using ProHema-CB following busulfan/cyclophosphamide/ATG conditioning for pediatric patients with inherited metabolic disorders.

A maximum of 12 eligible male and female subjects (1 to 18 years old, inclusive) will be enrolled and treated in the trial at approximately 1 to 3 centers within the U.S.

All subjects will be admitted to the hospital, per institutional practice and will receive a conditioning regimen, after which they will receive a HLA-matched or partially matched ProHema -CB unit on Day 0.

They will receive study follow up assessments weekly following Day 0 through Day 100 and study visit Days 180, 270, 365 and 730.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a confirmed diagnosis of an inherited metabolic disorder (IMD) and be amenable to treatment by hematopoietic cell transplantation:

   * Mucopolysaccharidoses: Hurler Syndrome (MPS IH), MPS I-HS (Hurler-Scheie Syndrome), Hunter Syndrome (MPS II), Sanfilippo Syndrome (MPS III), or MPS VI (Maroteaux-Lamy syndrome) with early neurologic involvement and/or sensitization to enzyme replacement therapy (ERT); or
   * Leukodystrophies: Krabbe disease (Globoid Leukodystrophy), Metachromatic Leukodystrophy (MLD), Adrenoleukodystrophy (ALD and AMN); or
   * Other IMD with lysosomal storage disorder including glycoproteinoses (Alpha-Mannosidosis, Mucolipidosis II or I-Cell disease), sphingo- and other lipidoses (Sandhoff disease, Tay Sachs disease, Pelizaeus Merzbacher (PMD), Niemann-Pick disease, GM1 gangliosidosis, Wolman's disease.
2. Male and female subjects aged 1 to 18 years, inclusive.
3. Lack of 4 6/6 HLA matched non-carrier related UCB or 8/8 HLA A, B, C, DRß1 matched non-carrier related or 8/8 unrelated bone marrow donor; or donor not available within appropriate timeframe, as determined by the transplant physician.
4. Availability of suitable primary and secondary umbilical cord blood (UCB) units.
5. Adequate performance status, defined as:

   * Subjects ≥ 16 years: Karnofsky score ≥ 70%.
   * Subjects < 16 years: Lansky score ≥ 70%.
6. Cardiac: Left ventricular ejection fraction at rest must be > 40%, or shortening fraction > 26%.
7. Pulmonary:

   * Subjects > 10 years: DLCO (diffusion capacity) > 50% of predicted (corrected for hemoglobin)
   * FEV1, FVC > 50% of predicted; Note: If unable to perform pulmonary tests, then O2 saturation > 92% on room air.
8. Renal: Serum creatinine within normal range for age, or if serum creatinine outside normal range for age, then renal function (creatinine clearance or GFR) > 70mL/min/1.73m2.
9. Hepatic: Bilirubin ≤ 2.5 mg/dL (except in the case of Gilbert's syndrome, ongoing hemolytic anemia, or due to the primary IMD); and ALT, AST and Alkaline Phosphatase ≤ x 3 ULN (all elevations beyond the ULN must be secondary to the primary IMD and not a comorbid condition).
10. Signed IRB approved Informed Consent Form (ICF).

Exclusion Criteria:

1. Evidence of HIV infection or HIV positive serology.
2. Current uncontrolled bacterial, viral or fungal infection (progression of clinical symptoms despite therapy).
3. Requirement for continuous respiratory supportive therapy (e.g. ventilator). Patients on intermittent respiratory support should be discussed with the Sponsor.
4. Active problems related to chronic aspiration.
5. Uncontrolled seizures.
6. Any active malignancy or myelodysplastic syndrome or any history of malignancy.
7. Inability to give informed consent/assent or to comply with the requirements for care after allogeneic stem cell transplantation.
8. Female subjects that are breastfeeding or with a positive pregnancy (HCG) test at Screening.
9. Use of an investigational drug within 30 days prior to screening for the primary IMD.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2015-06; Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Storgard, MD, Study Director — Fate Therapeutics
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ProHema-CB
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ProHema-CB
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] | 1.0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety Profile, Assessed Primarily by Neutrophil Engraftment
Time Frame: Engraftment by Day 42 following study transplant procedure
Measure: Count of Participants; unit: Participants
Arm/Group | ProHema-CB
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: During the First Year of Transplant
Description: Serious Adverse Events and Adverse Events assessed as possibly or probably related to ProHema are included below.
Arm/Group | ProHema-CB
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes